CLINICAL TRIAL: NCT03171909
Title: Austrian Registry on the Outcome of Monochorionic Multiple Pregnancies: A Multicenter Registry Study
Brief Title: Austrian Registry on the Outcome of Monochorionic Pregnancies
Acronym: MonoReg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other); Medical University Innsbruck (Other); Johannes Kepler University of Linz (Other); Paracelsus Medical University (Other); Klinikum Klagenfurt am Wörthersee (Other); Brothers of Saint John of God Eisenstadt (Unknown); SMZ-Ost Donauspital (Other); Hospital Hochsteiermark (Unknown); Landesklinikum Sankt Polten (Other); Klinikum Wels-Grieskirchen (Other); Landeskrankenhaus Feldkirch (Other); Landesklinkum Wiener Neustadt (Other); Mödling Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1497/2016
Record Dates: First submitted 2017-05-15; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Twin Dichorionic Diamniotic Placenta; Twin Monochorionic Monoamniotic Placenta; Twin-To-Twin Transfusion Syndrome; Twin Pregnancy With Antenatal Problem
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
About one third of twin pregnancies are resulting from a single fertilized oocyte. Two third of these monozygotic twins share a common placenta and are therefore called monochorionic. Due to placental sharing and the ever-present inter-fetal vascular connections, specific complications may arise and lead to an increased risk of intrauterine death and long-term neurodevelopmental impairment. Specific complications include twin-to-twin transfusion syndrome (TTTS), twin-anemia-polycythemia sequence (TAPS), selective intrauterine growth restriction (sIUGR) and discordant major anomalies, occurring in about 10%, 5%, 20% and 6% of monochorionic diamniotic twins. Prenatal interventions may improve perinatal and long-term outcome of affected fetuses. However, general knowledge about early diagnosis of monochorionic twins and their specific complications is still limited in a significant number of practitioners in Austria and systematic analysis of pregnancy outcomes are not conducted.

In this prospective multicenter registry study, the investigators aim to include all monochorionic pregnancies in Austria. Main outcome parameter is the occurrence of complications. Secondary outcomes are gestational age at occurrence of complications, gestational age delivery and neonatal outcome. The investigators also strive for long-term outcome, especially of infants following complicated pregnancies or preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* All monochorionic pregnancies diagnosed from 11+0 weeks of gestation

Exclusion Criteria:

* Dichorionic twin pregnancies or higher-grade multiples without a monochorionic pair

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All monochorionic pregnancies diagnosed from 11+0 weeks of gestation on
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of specific complications | from 12 weeks of gestation to delivery
  TTTS, sIUGR, TAPS, TRAP, IUFD, malformations, miscarriage

SECONDARY OUTCOMES:
gestational age at delivery | at delivery
  gestational age (weeks+days) at delivery
birth weight | at first day of life
  birth weight in grams
body length at birth | at first day of life
  body length in cm
umbilical artery pH-value | immediately after birth
  pH-Value derived from umbilical cord blood after birth
cord blood hemoglobin levels | immediately after birth
  hemoglobin levels derived from umbilical cord blood after birth
APGAR score | within 10 min after birth
  APGAR score 1, 5 and 10 min following delivery
neonatal complications | within 1 month after birth
  occurrence of neonatal complications including neonatal death, cerebral hemorrhage, periventricular leucomalacia, bronchopulmonary dysplasia, sepsis, retinopathy of the newborn, necrotizing enterocolitis, seizures
long-term outcome | 2 years of age
  Neurodevelopmental outcome should be performed at the corrected age of 2 years. If available, neurodevelopment will be assessed by using the Bayley Scales of Infant Development. In other cases the Bayleys or the Ages & Stages Questionnaires may be used.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Klaritsch, MD, Principal Investigator — Department of Obstetrics and Gynecology, Medical University of Graz, Austria
Locations (13):
- Austria (13):
  - Medical University of Graz, Graz, Styria
  - Brothers of Saint John of God Eisenstadt, Eisenstadt
  - Medical University Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Hospital Hochsteiermark, Leoben
  - Johannes Kepler University of Linz, Linz
  - Mödling Hospital, Mödling
  - Paracelsus Medical University, Salzburg
  - Landesklinikum Sankt Polten, Sankt Pölten
  - Medical University Vienna, Vienna
  - SMZ-Ost Donauspital, Vienna
  - Klinikum Wels-Grieskirchen, Wels
  - Klinikum Wiener Neustadt, Wiener Neustadt

IPD SHARING:
Plan to Share IPD: No